CLINICAL TRIAL: NCT05533762
Title: The Effect of Insoles on Functional Performance in Pediatric Flexible Flatfoot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: N202106064
Record Dates: First submitted 2022-08-11; First posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-08

CONDITIONS: Flatfoot, Flexible
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arch insole (Active Comparator): Half of the subjects are randomly assigned to assess balance capacity with arch insole first.
  Three day wash out, the subjects are assess balance capacity with sham insole.
  Interventions: Device: arch insole and sham insole
- sham insole (Sham Comparator): Half of the subjects are randomly assigned to assess balance capacity with sham insole first.
  Three day wash out, the subjects are assess balance capacity with arch insole.
  Interventions: Device: arch insole and sham insole

INTERVENTIONS:
Device: arch insole and sham insole — children wear insoles on feet

SUMMARY:
Flexible flatfoot is a condition that increase the load of the foot structure.With prolonged standing or walking, some children with flatfoot experience rapid discomfort or fatigue in the foot In this study, the investigators investigated the short-term effects of customized insoles on body functions and structures, and activities and participation in children with flexible flatfoot.

DETAILED DESCRIPTION:
Flexible flatfoot is a condition that involves the collapse of the medial longitudinal arch of the foot during weight-bearing stress and the restoration of the arch after the removal of body weight.

Flatfoot may increase the load of the foot structure, potentially interfering with normal foot function. With prolonged standing or walking, some children with flatfoot experience rapid discomfort or fatigue in the foot, pain in the plantar foot, and instability of the medial foot structure. Treatment effect of corrective shoes or insoles on flexible flatfoot in children remain uncertain.

In this study, the investigators investigated the short-term effects of customized insoles on body functions and structures, and activities and participation in children with flexible flatfoot. The investigators hypothesized that the short-term use of customized insoles improves the scores for measures of body functions and structures and activities and participation.

The investigators hypothesized that the short-term use of customized insoles improves the scores for measures of body functions and structures and activities and participation.

ELIGIBILITY:
Inclusion Criteria:

* Children presenting symptomatic flexible flatfoot only

Exclusion Criteria:

* Children with a history of foot injury or surgery, foot abnormalities or a confirmed diagnosis such as neurological deficits.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Functional Reach Test(FRT) from pre to post-intervention. | up to 10 minutes
  The Functional Reach Test (FRT) is a quick screen for determining balance capacity.
Pediatric Berg Balance Scale | up to 30 minutes
  Pediatric Berg Balance Scale was developed to measure balance among older people with impairment in balance function by assessing the performance of functional tasks.
  Maximum score is 56 ,and minimum values is 0. Score 54-56 means a better outcome.

SECONDARY OUTCOMES:
Change in Center of pressure (CoP) from pre to post-intervention. | up to 30 minutes
  The center of pressure (CoP) measures derived from the foot pressure mat and force plate of RSSCAN system.

CONTACTS AND LOCATIONS:
Overall Officials: YenTing LIU, Master, Study Chair — Wang Fang Hospital, Taipei Medical University

IPD SHARING:
Plan to Share IPD: No